CLINICAL TRIAL: NCT06360536
Title: Remotely Delivered Resistance Training for Cardiometabolic Health Among Black Women: A Pilot Trial
Brief Title: Remotely Delivered Resistance Training for Cardiometabolic Health Among Black Women
Acronym: OVERCOME-IT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Amber W. Kinsey, PhD, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300012634; P50MD017338 (NIH)
Record Dates: First submitted 2024-04-04; First posted 2024-04-11 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Overweight or Obesity; Prediabetes or Diabetes; Prehypertension (Elevated Blood Pressure) or Hypertension; Resistance Training
MeSH Terms: conditions — Overweight; Obesity; Prediabetic State; Diabetes Mellitus; Prehypertension; Hypertension | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention/Treatment (Experimental): A home-based resistance training condition that is delivered through a web-based platform.
  Interventions: Behavioral: Resistance Training

INTERVENTIONS:
Behavioral: Resistance Training — A home-based resistance training condition that is delivered through a web-based platform.
  Other Names: RT

SUMMARY:
The purpose of this study is to collect preliminary data on the feasibility, acceptability, and potential effects of a novel, remotely delivered resistance training program.

DETAILED DESCRIPTION:
This trial will enroll Black women with elevated cardiometabolic risk (e.g., overweight or obesity, pre- or established diabetes, and elevated or high blood pressure) in early-to-middle adulthood (n=36; age=30-64 years) with insufficient resistance training (RT) participation. This 4-month single group pilot trial evaluates the feasibility, acceptability, and potential effects of a novel, remotely-delivered resistance training (RT) intervention. All participants will engage in RT during this trial and the web-based platform is the primary modality through which the remote RT intervention is delivered. Assessments are conducted at baseline and follow-up (month 4). Aim 1 will examine the feasibility and acceptability of the remotely delivered RT program. Aim 2 will examine the potential effects on RT behaviors. Aim 3 will examine the potential effects on clinical and patient-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Self-identifies as Black or African American
* Female
* Age 30-64 years
* Insufficient resistance training engagement (<2 sessions/week in the past 6 months)

AND

* Self-reported or documented diagnosis of at least one of the following conditions: Overweight, obesity, prediabetes, type 2 diabetes, elevated blood pressure, hypertension, or taking medications for any of these conditions
* Has an internet- connected device (i.e., computer, smartphone) and is willing to use it for intervention delivery
* If indicated during screening, willing to obtain medical clearance for exercise from their healthcare provider prior to enrollment
* Residing within a 50-mile radius of the University

Exclusion Criteria:

* Uncontrolled hypertension (blood pressure >160/100 mm Hg)
* Weighing ≥ 450 lbs (upper limit for body composition assessment)
* Conditions or limitations that affect physical activity participation and/or the ability to --perform assessments
* Has a medical or physical condition that make moderate intensity physical activity (like a brisk walk) difficult or unsafe
* Unwilling to obtain medical clearance (if indicated by prescreening)
* Women who are pregnant or trying to become pregnant in the next 6 months
* Planning to relocate out of the area in the next 6 months
* Participating in another exercise and/or randomized research project
* Unwilling or unable to do any of the following: give informed consent; read/understand English; perform resistance training in their home, record and upload virtual exercise assessment sessions, and other protocol specific requirements

Ages: 30 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment | Baseline
  The number of participants enrolled in the trial
Feasibility of retention | Month 4
  The proportion of participants who complete the study out of those who enrolled in the study
Intervention adherence | Month 4
  The number of participants adhering to the intervention

SECONDARY OUTCOMES:
Change in resistance training behaviors | Baseline and Month 4
  The number of days of resistance training completed
Change in blood pressure | Baseline, Month 4
  Systolic and diastolic blood pressure measured by an automated device
Change in HbA1C | Baseline, Month 4
  HbA1C measured by a point-of-care device
Change in body composition | Baseline, Month 4
  Percent body fat measured by dual-energy x-ray absorptiometry
Change in handgrip strength | Baseline, Month 4
  The highest value of 3 maximal attempts on each hand
Change in the number of chair stands | Baseline, Month 4
  The number of chair stands completed in 30 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Amber W Kinsey, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States